CLINICAL TRIAL: NCT04260178
Title: The Impact Of An Education-Based Intervention Program (EBIP) On Dyspnea And Chronic Self-Care Management Among Copd Patients: A Randomized Controlled Study
Brief Title: Education-Based İntervention Program for Persons With Chronic Obstructive Pulmonary Disease (EBIPCOPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gönül GÖKÇAY (Other)
Responsible Party: Sponsor-Investigator, Gönül GÖKÇAY, Lecturer, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 80576354-050-99/37
Record Dates: First submitted 2020-01-24; First posted 2020-02-07 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; dyspnea; self-care management; nurse education.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Hospitals; Home Care Services; Body Mass Index

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Double blinding is not considered possible for EBIP interventions, where participants and researcher can recognize group assignment. However, giving and scoring the assessments were masked wherever feasible. The assistant researcher who administered and scored the questionnaires and the nurse that carried out PFT measurement and assessments were blind to experimental groups. Coded answer sheets were analyzed only after the study's completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental groups (Experimental): For the experimental group, EBIP was implemented in three stages:(1) hospital training;(2) home visits + training, which includes motivational interventions that facilitate chronic disease self-care and symptom management with nurse-patient cooperation; and (3) telephone follow-ups and assistance. A handbook was developed in line with the relevant literature and input from two specialist physicians (1,17-20). The handbook consisted of 4 sections that concerned improving breathing exercises, drug compliance, nutrition and illness self-care behavior. The trainings sessions were conducted in a hospital seminar room using PowerPoint presentations. Afterward, patients were asked to demonstrate what they learned, and the parts that were not clear were explained again. The training was concluded after deciding for the first home visit appointment. For patients that could not effectively use the handbook, a close relative was included to all steps of the study.
  Interventions: Other: An Education-Based Intervention Program and handbook (EBIP, hospital and home); Other: PFT, BMI, BDI, SCMP-G
- Control groups (Other): Control groups were evaluated with an introductory survey form, PFT, BDI, BMI and SCMP-G scales before and after the study. There were no additional interventions to the control group.
  Interventions: Other: PFT, BMI, BDI, SCMP-G

INTERVENTIONS:
Other: An Education-Based Intervention Program and handbook (EBIP, hospital and home) — A handbook was developed in line with the literature and input from two specialist physicians. The handbook consisted of 4 sections that concerned improving breathing exercises, drug compliance, nutrition and illness self-care behavior.
  Arms: Experimental groups
Other: PFT, BMI, BDI, SCMP-G — pulmonary function test(PFT), the Baseline Dyspnea Index(BDI), body mass index(BMI) and the Self Care Management Process in Chronic Illness(SCMP-G) scale

SUMMARY:
Obstructive Pulmonary Disease(COPD) treatment, leading to the role of nurses to become more and more important. An Education-Based Intervention Program(EBIP) consists of several steps that aim to achieve better health outcomes through guidingCOPD patients to reduce dyspnea symptoms and improve chronic self-care management skills. The aim of this study is to evaluate the dyspnea and chronic self-care management outcomes of EBIP compared to routine care.

Research Hypotheses:

H0: EBIP has no effect on dyspnea or chronic self-care management in COPD patients.

H1: EBIP effects dyspnea outcomes of COPD patients. H2: EBIP effects chronic self-care management outcomes of COPD patients.

DETAILED DESCRIPTION:
Abstract:

Background:Non-pharmacological interventions are a valuable aspect of Chronic Obstructive Pulmonary Disease(COPD) treatment, leading to the role of nurses to become more and more important. An Education-Based Intervention Program(EBIP) consists of several steps that aim to achieve better health outcomes through guidingCOPD patients to reduce dyspnea symptoms and improve chronic self-care management skills. The aim of this study is to evaluate the dyspnea and chronic self-care management outcomes of EBIP compared to routine care.

Method:A total of 61 Stage II COPD patients that were hospitalized and treated in the month of January 2019 in a university hospital were selected for the study, who had been discharged less than one month ago and resided downtown. 51 conforming patients were divided into experimental(EBIP intervention) and control groups for a single-blind randomized trial. Data were collected using an introductory information form, pulmonary function test(PFT), the Baseline Dyspnea Index(BDI), body mass index(BMI) and the Self Care Management Process in Chronic Illness(SCMP-G) scale. There were no addition interventions to the control group. The intervention group underwent a 3-month EBIP intervention that included education, house visits and follow-ups through phone calls. The data were analyzed using SPSS version 17.0 with descriptive statistics, x2,Mann Whitney U and Wilcoxon signed-rank tests. p<0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals to be included in the study are 18 years of age and over
* have been diagnosed with COPD Stage 2 for six months or more,
* not having been in hospital for one month after discharge, - no communication problems,
* lack of mental confusion,
* conscious and complete orientation
* volunteering to participate in the research,
* It is planned to be conducted with patients living in the center of Kars.

Exclusion Criteria:

* Being 18 years old and under,
* KOAH stage 1, 2, 4 diagnosed,
* being a communication problem,
* having mental confusion or
* having any psychiatric problem,
* not volunteering to participate in the research,
* Living outside the Kars center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
pulmonary function test(PFT) | Change from PFT at 3 months
  It is the COPD diagnostic criterion that the ratio of these two values is below 70% by measuring the forced vital capacity (FVC) with PFT and the demanding expiration volume (FEV1) in the first second and the ratio of these two values is calculated by FEV1 / FVC (% FEV1 predicted). According to the GOLD 2019 classification; 1. Stage-mild (FEV1≥80% predicted), 2. Stage-moderate (50% ≤FEV1 <80% predicted), 3. Stage-severe (30% ≤FEV1 <50% predicted), 4. Stage-very severe ( FEV1 <30% predicted). In our study, the changes in FVC, FEV1, FEV1 / FVC (% FEV1) values were measured by including 2nd stage COPD patients.
Baseline Dyspnea Index(BDI) | Change from BDI at 3 months
  The BDI score is based on ratings for three categories: functional impairment, size of task, and extent of effort. Dyspnea in each category is rated on a 5-point scale from 0 (severe) to 4 (intact). The scores of each category are added to create a total dyspnea score (between 0 and 12). Higher scores indicate worse dyspnea.
Self-Care Management Scale in Chronic Diseases(SCMP-G) | Change from SCMP-G at 3 months
  Scale with 35 questions; These two types of protection concepts, defined as self-protection (20 items) and social protection (15 items), constituted two sub-dimensions of the scale. Self-protection sub-dimension items 2, 6, 8, 11, 15, 18, 19, 20, 22, 23 and 25-34 and social-protection sub-dimension 1, 3-5, 7, 9, 10, 12-14, 16 Consists of 17, 21, 24 and 35 items. The assessment of the scale was developed from a 5-point Likert form as 5 (Strongly Agree) and 1 (Never Agree). Questions 3, 15, 19, and 28 on the SCMP-G scale are in the form of a negative question and the evaluation needs to be transformed. Self-care management increases as the score on the SCMP-G scale increases.The overall Cronbach alpha values of the scale are 0.75, 0.78 for the self-protection sub-dimension and 0.78 for the social-protection sub-dimension.

SECONDARY OUTCOMES:
body mass index(BMI) | Change from BMI at 3 months
  BMI was measured using weight and height data. Height was measured with a stadiometer (precision 1 cm) and weight was measured using a standard medical weighing scale (precision 1 kg). The interview was concluded for the control group at this point.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ÇEVİRME, Principal Investigator — Sakarya University
Locations (2):
- Turkey (Türkiye) (2):
  - Sakarya University Health Faculty of Health Sciences, Sakarya, Turke/Sakarya
  - Kafkas University-Ataturk Health Services Vocational School, Kars, Turkey/Kars

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thom DH, Willard-Grace R, Tsao S, Hessler D, Huang B, DeVore D, Chirinos C, Wolf J, Donesky D, Garvey C, Su G. Randomized Controlled Trial of Health Coaching for Vulnerable Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2018 Oct;15(10):1159-1168. doi: 10.1513/AnnalsATS.201806-365OC. PMID 30130430
- [Result] Baker E, Fatoye F. Patient perceived impact of nurse-led self-management interventions for COPD: A systematic review of qualitative research. Int J Nurs Stud. 2019 Mar;91:22-34. doi: 10.1016/j.ijnurstu.2018.12.004. Epub 2018 Dec 31. PMID 30669076
- [Result] Efraimsson EO, Hillervik C, Ehrenberg A. Effects of COPD self-care management education at a nurse-led primary health care clinic. Scand J Caring Sci. 2008 Jun;22(2):178-85. doi: 10.1111/j.1471-6712.2007.00510.x. PMID 18489687
- See also: Global Inıtıatıve For Chronıc Obstructıve Lung Dısease. Pocket Guıde To Copd Dıagnosıs, Management, And Preventıon. — https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-POCKET-GUIDE-FINAL_WMS.pdf